CLINICAL TRIAL: NCT04029272
Title: Study on the Effect of Metformin vs Metformin Combined With GLP-1 RA (Exenatide) on Overweight/Obese Patients With Polycystic Ovary Syndrome (PCOS)
Brief Title: Metformin vs Metformin Combined With GLP-1RA (Glucagon-like Peptide 1 Receptor Agonist) on Overweight/Obese PCOS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Aijun Sun, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS201907
Record Dates: First submitted 2019-07-08; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; GLP-1; GLP-1RA; exenatide; Metformin; glucagon-like peptide 1; glucagon-like peptide 1 receptor agonist
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Background therapy: Diane-35 one pill by mouth, once daily, beginning on Day 5 of the menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles (3 months)
  Metformin: Metformin was initiated at a dose of 250mg q.d. and increased by 250mg up to 500 mg t.i.d.
  Interventions: Drug: Metformin
- Metformin+EQW (Experimental): Background therapy: Diane-35 one pill by mouth, once daily, beginning on Day 5 of the menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles (3 months)
  Metformin: Metformin was initiated at a dose of 250mg q.d. and increased by 250mg up to 500 mg t.i.d.
  EQW: Participants will receive long-acting Exenatide once a week for 12 weeks
  Interventions: Drug: Metformin; Drug: Exenatide 2 MG

INTERVENTIONS:
Drug: Metformin — 500 mg tid for 12 weeks
  Other Names: Glucophage
Drug: Exenatide 2 MG — Exenatide injection once weekly for 12 weeks
  Other Names: Bydureon
  Arms: Metformin+EQW

SUMMARY:
The purpose of this study was to determine whether metformin combined with exenatide once weekly (EQW) is more effective than metformin alone in the treatment of overweight/obese women with polycystic ovary syndrome (PCOS). Background therapies were Diane-35 or/and progesterone capsule. 80 participants were randomized to use either metformin or metformin+EQW for 12 weeks. Greater changes in body weight were anticipated in patients treated with EQW+metformin than metformin alone in those treated with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years to 40 years of age
* Diagnosed as PCOS by the 2003 Rotterdam criteria.
* Overweight/obesity (BMI≥25 kg/m2)
* No pregnant plan in recent 6 months
* Written consent for participation in the study

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* Subjects have other endocrine diseases, such as adrenal hyperplasias or tumor, androgen-secreting tumors, Cushing's syndrome, thyroid diseases, and hyperprolactinemia
* Diagnosed with or have a family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* Serious systemic disease or malignant tumor
* History of pancreatitis (chronic, acute or recurrent)
* Body weight change ≥10% at 3 months before treatment
* Used oral contraceptives or sex hormone drugs in the past 1 month
* Used oral glucocorticoids in the past 1 month
* Substance (alcohol or drug) abuse or dependence within 3 months; Heavy smokers (smokers who smoke 20 or more cigarettes a day) or heavy drinkers (>10g/d)
* Subjects have a severe systemic disease, such as cardiovascular system
* Renal impairment, eGFR<60ml/min/1.73m2
* Increase of transaminases up to < 2.5 times of upper limit of normal value
* Have a history of thromboembolic disease or thrombotic tendency
* Subjects in pregnant or lactating or within 1 year after delivery.
* Subjects have an allergic history to the drugs used in the study
* Subjects have participated in other clinical researches of medicine within 1 month prior to randomization.
* Use of metformin, glucagon-like peptide -1 receptor agonists, or weight loss medications (prescription or OTC) within 30 days before screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Patient's body weight was measured at the baseline and after 12 weeks of clinical trial

SECONDARY OUTCOMES:
Proportion of subjects who lost ≥5% of their body weight | 12 weeks
Proportion of subjects who lost ≥ 10% of their body weight | 12 weeks
Change in body mass index (BMI) | 12 weeks
Change in waist circumference(WC) | 12 weeks
Change in hip circumference (HC) | 12 weeks
Changes in lipid accumulation product(LAP) | 12 weeks
  LAP=(WC(cm)-58)×TG (mmol/L)
Changes in Visceral obesity index(VAI) | 12 weeks
  VAI = (WC(cm)/39.68+(1.88×BMI))×(TG (mmol/l)/1.03)×(1.31/HDL (mmol/l))
Changes in blood pressure | 12 weeks
Changes in Blood Glucose and Insulin During the oral glucose tolerance test (OGTT) | 12 weeks
  glucose obtained at 0,30,60 and 120 minutes during the OGTT. HOMA-IR=Glu0(mmol/l)×Ins0(mU/ml)/22.5
  Matsuda index=1000/ square(Ins0 (mU/ml) ×Glu0 (mmol/l)×mean Glu(mmol/l)×meanIns(mU/ml)]
  QUICKI= 1/Log[Glu0 (mU/ml) ×Ins0 (mmol/l)]
  HOMA-β=20×Ins0 (mU/ml) /(Glu0 (mmol/l)-3.5)
  MBCI= Ins0 (mU/ml)×Glu0(mmol/l)／(Glu120(mmol/l)＋Glu60 (mmol/l)-2×Glu0 (mmol/l)）
  ΔI30/ΔG30 = (Ins30- Ins0)/( Glu30- Glu0)
Changes in total cholesterol (TC) | 12 weeks
Changes in serum triglyceride (TG) | 12 weeks
Changes in high-density lipoproteincholesterol (HDL-C) | 12 weeks
Changes in low-density lipoproteincholesterol (LDL-C) | 12 weeks
Changes in lipoprotein(a) | 12 weeks
Changes in apolipoprotein a1(ApoA1) | 12 weeks
Changes in apolipoprotein B(ApoB) | 12 weeks
Changes in free fatty acid (FFA) | 12 weeks
Changes in high sensitivity C reactive protein(hsCRP) | 12 weeks
Frequency of menstrual cycle | 12 weeks
  The number of menstrual cycles during the previous year was recorded and the menstrual cycle ratio calculated by dividing 12 by the number of menstrual cycles in the previous year . During the study period, the patients in a menstrual diary recorded vaginal bleeding over 12 weeks. The effects of treatment intervention on menstrual cycle interval was calculated evaluated by dividing 3 by the number of menstrual cycles recorded in each patient's menstrual cycle diary.
Changes in testosterone | 12 weeks
Changes in Dehydroepiandrosterone sulfate (DHEAS) | 12 weeks
Changes in Luteinizing Hormone (LH) | 12 weeks
Changes in follicle stimulating hormone(FSH) | 12 weeks
Changes in LH/FSH | 12 weeks
Changes in Acne severity score | 12 weeks
  This system divides the face, chest, and upper back into 6 areas: the forehead, right cheek,left cheek, nose, chin, and torso (chest and upper back combined). Each acne lesion is described and scored as a comedo (1 point), papule (2 points), pustule (3 points), or nodule (4 points); absence of an acne lesion in an area results in a score of 0 points. The local score for each anatomic area is determined by multiplying the score of the most severe lesion by an area factor (1 to 3), and the local scores of the 6 areas are then added together to obtain the total score. Acne severity is graded as none (total score, 0 points), mild (total score, 1-18 points), moderate (total score, 19-30 points), severe (total score, 31-38 points), and very severe (total score N38 points)
Changes in ovarian volume | 12 weeks
Changes in follicular number of 2-9mm in diameter | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xuesong D, Tao T, Weilu W, Wei X, Wei X, Yan D, Yanfang W, Ruilin M, Yingying G, Yue W, Perez-Lopez FR, Yang W. Combined metformin and exenatide versus only metformin treatments in polycystic ovary syndrome with abdominal obesity and network pharmacology of gene expression: evidence from a randomized clinical trial. Ther Adv Endocrinol Metab. 2025 Aug 19;16:20420188251355411. doi: 10.1177/20420188251355411. eCollection 2025. PMID 40843067
- [Derived] Ma RL, Deng Y, Wang YF, Zhu SY, Ding XS, Sun AJ. Short-term combined treatment with exenatide and metformin for overweight/obese women with polycystic ovary syndrome. Chin Med J (Engl). 2021 Nov 3;134(23):2882-2889. doi: 10.1097/CM9.0000000000001712. PMID 34732660